CLINICAL TRIAL: NCT02657512
Title: Effect of Activated Charcoal on Rivaroxaban Pharmacokinetics in Healthy Subjects : RICHAR Study
Brief Title: Effect of Activated Charcoal on Rivaroxaban Pharmacokinetics in Healthy Subjects
Acronym: RICHAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 1508030; 2015-001839-21 (EudraCT Number); 140096A-21 (Other: ANSM)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Rivaroxaban, pharmacokinetics, activated charcoal, poisoning
MeSH Terms: conditions — Anthrax; Poisoning | interventions — Rivaroxaban; Charcoal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): * Period " rivaroxaban alone"
  * Washout period (at least 6 days)
  * Period " rivaroxaban and activated charcoal 2 hours after rivaroxaban administration"
  * Washout period (at least 6 days)
  * Period " " rivaroxaban and activated charcoal 5 hours after rivaroxaban administration"
  Interventions: Drug: rivaroxaban; Drug: rivaroxaban and activated charcoal
- Arm B (Experimental): . Period " rivaroxaban and activated charcoal 5 hours after rivaroxaban administration"
  * Washout period (at least 6 days)
  * Period " rivaroxaban alone"
  * Washout period (at least 6 days)
  * Period " " rivaroxaban and activated charcoal 8 hours after rivaroxaban administration"
  Interventions: Drug: rivaroxaban; Drug: rivaroxaban and activated charcoal
- Arm C (Experimental): . Period " rivaroxaban and activated charcoal 2 hours after rivaroxaban administration"
  * Washout period (at least 6 days)
  * Period " " rivaroxaban and activated charcoal 8 hours after rivaroxaban administration"
  * Washout period (at least 6 days)
  * Period " rivaroxaban alone"
  Interventions: Drug: rivaroxaban; Drug: rivaroxaban and activated charcoal

INTERVENTIONS:
Drug: rivaroxaban — rivaroxaban 40 mg/day (1 day)
Drug: rivaroxaban and activated charcoal — rivaroxaban 40 mg/day (1 day) and 50 g of activated charcoal 2 or 5 or 8 hours after rivaroxaban administration (1 day)

SUMMARY:
Rivaroxaban is a direct oral anticoagulant that target specifically activated factor X. Bleeding events related to rivaroxaban are the consequence of physiopathologic, pharmacokinetic issues or poisoning. Few results are available on the use of activated charcoal in rivaroxaban poisoning. Moreover, a recent study, in healthy subjects, shows that activated charcoal can reduce significantly exposition to apixaban (a direct oral anticoagulant of the same class). The objective of this study is to evaluate the effect of activated charcoal on rivaroxaban pharmacokinetics. It corresponds to a randomised open trial with an incomplete cross over design (3 occasions). It will enrol 12 healthy subjects. Four treatments modalities will be studied: rivaroxaban alone and rivaroxaban with activated charcoal administrated 2, 4 or 8 hours after rivaroxaban administration.

ELIGIBILITY:
Inclusion Criteria:

* affiliated or beneficiary of a social security category
* having signed the inform consent form
* having signed the genetic consent form
* BMI between 18.5 and 25
* normal clinical exam
* normal biological exam

Exclusion Criteria:

* contra-indication to rivaroxaban
* contra-indication to activated charcoal
* previous history of psychiatric disease, or antidepressant treatment, or convulsion, or hemorrhagic disease smoker
* Organic lesion likely to bleed
* severe liver disease
* severe kidney failure
* previous surgery within one month

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of rivaroxaban | H0.5, H0.75, H1, H1.5, H2, H2.5, H3, H4, H5, H6, H8, H10, H12, H14, H18 and H24 after rivaroxaban administration
  rivaroxaban pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ollier E, Hodin S, Lanoiselee J, Escal J, Accassat S, De Magalhaes E, Basset T, Bertoletti L, Mismetti P, Delavenne X. Effect of Activated Charcoal on Rivaroxaban Complex Absorption. Clin Pharmacokinet. 2017 Jul;56(7):793-801. doi: 10.1007/s40262-016-0485-1. PMID 27910037